CLINICAL TRIAL: NCT00760695
Title: Cannabinoid CB1 Receptor Agonist Treatment in Severe Chronic Anorexia Nervosa
Brief Title: Cannabinoid Receptor (CB1) Agonist Treatment in Severe Chronic Anorexia Nervosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Tine Hylle, for Alin Andries, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 033
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; chronic; dronabinol; weight gain; EDI
MeSH Terms: conditions — Anorexia Nervosa; Bronchiolitis Obliterans Syndrome; Weight Gain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): the patients in this arm are receiving 2,5 mg dronabinol twice daily
  Interventions: Drug: dronabinol
- B (Placebo Comparator): the patients in this arm are receiving 2,5 mg placebo twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dronabinol — tablets, twice daily, for 4 weeks
  Other Names: Marinol
  Arms: A
Drug: placebo — tablets, twice daily, for 4 weeks
  Arms: B

SUMMARY:
A pilot study designed to reveal the effects of Marinol / dronabinol, a CB 1 agonist.

Primary end point: To estimate weight gain and EDI scores in patients receiving Marinol compared to placebo

Secondary end points: Motor and inner restlessness and hormonal changes during the treatment.

DETAILED DESCRIPTION:
The goals of this study are to reveal through a pilot trial if treatment of patients with severe chronic AN with Marinol® (dronabinol, a CB1 agonist) has significant effect on:

* Weight
* Eating Disorder Inventory (EDI) scale
* Motor and inner restlessness (estimated by accelerometry)
* Endocrine parameters (see below, paragraph 4.4) This study is a randomized, double blinded, placebo controlled cross over study. 24 patients with chronic AN meeting the inclusion criteria will be randomized either to receive Marinol® or placebo. After four weeks the two groups will undergo a wash-out period and after that will receive the opposite therapeutic regime for another four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients under treatment for AN.
* Patients attending ambulatory treatment, which are not expected to be admitted at the hospital with AN-related pathology or discharged during the study period.
* Patients admitted to Department of Endocrinology M or Psychiatric Department P which are not expected to be discharged during the study period.
* Age over 18.
* Duration of the disease over 5 years.

Exclusion Criteria:

* Patients under compulsory treatment or suffering of mania, schizophrenia or primary depression.
* Patients with any medical or psychiatric event related or not related to the underlying eating disorder which requires prolonged admission to the hospital during the study.
* Patients with unstable heart disease (relevant changes in medication prior or during the study) and limitation of activity (not comfortable with more than moderate exertion / at rest).
* Patients not attending to the weekly controls.
* If other severe adverse events (SAE) / drug reactions (SADR) are suspected.
* Patients actually having or having a history of alcohol, cannabis, opioids or central stimulating drugs abuse.
* Patients with known allergy to dronabinol or sesame oil.
* Fertile, menstruating women not using safe contraception.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Weight gain | 4 weeks

SECONDARY OUTCOMES:
Eating Disorder Inventory (EDI) scale | 4 weeks
Motor and inner restlessness (estimated by accelerometry) | 4 weeks
Endocrine parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andries Alin, physician, Principal Investigator — Endocrinological Department, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark